CLINICAL TRIAL: NCT05370274
Title: Cranial Nerve Non-invasive Neuromodulation to Improve Pain and Upper Extremity Function in Individuals in the Chronic Phase of Stroke: a Pilot Feasibility Study
Brief Title: Using Cranial Nerve Non-invasive Neuromodulation to Improve Pain and Upper Extremity Function After a Stroke
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Université de Sherbrooke (Other)
Responsible Party: Principal Investigator, Marie-Hélène Milot, Principal Investigator, Université de Sherbrooke
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2022-4609
Record Dates: First submitted 2022-04-27; First posted 2022-05-11 (Actual); Last update posted 2024-02-23 (Actual); Status verified 2024-02

CONDITIONS: Stroke
Keywords: Exercise; Upper limb; Motor recovery; Pain; Cranial nerve non-invasive neuromodulation
MeSH Terms: conditions — Stroke; Motor Activity; Pain

STUDY DESIGN:
Intervention Model Description: The study model is a pre/post intervention pilot study.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- strength training intervention (Experimental): Strength training of the affected upper limb in chronic stroke survivors
  Interventions: Procedure: Strength training intervention
- Cranial nerve non-invasive neuromodulation (CN-NINM) (Experimental): CN-NINM will be applied during each session of the strength training intervention
  Interventions: Procedure: Cranial nerve non-invasive neuromodulation (CN-NINM)

INTERVENTIONS:
Procedure: Strength training intervention — The strength training program will last 4 weeks (3 X/week, 60 minutes). Using dead weights, the 1RM (i.e. the maximal load that an individual can lift once) will be estimated by the 10RM in order to avoid tendino-muscular injuries and fatigue. The 10RM will be determined for the muscles playing a key role in the functional performance of the upper limb (the wrist extensors and the elbow and shoulder flexors). In addition, the grip muscles of the affected hand will be trained with a JAMAR® dynamometer. Training will start at 50% of 1RM and progress by 10% each week to reach 80% of 1RM by week 4. The same gradation of intensity will be applied to the grip muscles. The training will begin and end by a 5-minute warm-up and relaxation period comprising of active movements of the trained muscles.
  Arms: strength training intervention
Procedure: Cranial nerve non-invasive neuromodulation (CN-NINM) — During each strength training session, the CN-NINM will be applied, with the help of a portable stimulator comprising a network of 18 electrodes, directly on the tongue of the participants for 20 minutes. The participants will hold the CN-NINM in place by pressing their tongue upwards. The CN-NINM will generate high-frequency pulses (50 μsec to 150 Hz), and the intensity of the stimulus will be set by each participant to a comfortable level of sensation, similar to the sensation in the mouth of a soft drink.
  Arms: Cranial nerve non-invasive neuromodulation (CN-NINM)

SUMMARY:
Following a stroke, individuals experience pain in the affected upper limb (UL) and residual weakness in the UL, which impacts their quality of life and performance of activities of daily living. To overcome these deficits, exercises are a key element to any rehabilitation program and are based on the reorganization capacity of the central nervous system (called neuroplasticity). To optimize the beneficial effects of exercises and potentiate neuroplasticity, non-invasive brain stimulation devices (NIBS) are increasingly used as a complementary therapy post stroke. Among NIBS, a new technique, called cranial nerve non-invasive neuromodulation (CN-NINM), is making its way into stroke rehabilitation since, unlike other NIBS such as tDCS, it allows the generation of a direct flow of neuronal impulses via the stimulation of the tongue. The goal of this project is therefore to investigate CN-NINM to document its feasibility and explore its efficacy at improving motor recovery and reduce pain at the affected UL in chronic stroke patients (> 6 months). CN-NINM will be applied for 20 minutes during each exercise session of the UL (3X/week, 4 weeks). Feasibility data will comprise adherence to CN-NINM, drop out rate and adverse events and UL motor recovery and pain will be assessed before and after the exercise program. At the end of this study, it is expected that it will be feasible to use CN-NINM as an intervention in combination with the exercise program and that it will result in improved motor function and reduced pain in affected UL.

DETAILED DESCRIPTION:
Following a stroke, survivors experience pain in the affected upper limb (UL) and residual weakness in the UL, which impacts their quality of life and performance of activities of daily living. Exercises is a key element of any rehabilitation program and is based on the capacity of reorganization of the central nervous system (called neuroplasticity) to allow overcoming stroke deficits. In addition, it is now recognized that in the chronic phase of a stroke, motor and functional gains are still possible following various training programs, such as a strength training program. To optimize the beneficial effects of exercise and potentiate neuroplasticity, non-invasive brain stimulation (NIBS) devices are increasingly used as a complementary therapy. Among NIBS, the most widely used technique is transcranial direct current stimulation (tDCS) that modulates cortical excitability and allows for clinical and functional gains, including recovering in UL motor function and pain. However, over 50% of individuals do not respond as expected to the combination of tDCS and rehabilitation exercises. This can be due to anatomical variability between individuals and electrical current shunting. Thus, to bypass these constraints, a new technique, called cranial nerve non-invasive neuromodulation (CN-NINM), is entering stroke rehabilitation. Unlike other NIBS such as tDCS, it generates a direct flow of neural impulses via tongue stimulation. Studies have shown that priming the motor cortex with CN-NINM during a training program can promote improved balance and gait and increased activation of the motor cortex. Until now, no studies have examined the use of CN-NINM for improving UL function and pain.

Goals: 1) To assess the feasibility of using CN-NINM in chronic stroke survivors; 2) To explore the effectiveness of CN-NINM in improving motor function and reducing pain of the affected upper limb in chronic stroke survivors.

Methods: In this feasibility pilot pre/post intervention study, 12 adults at the chronic phase of a stroke (>6 months) will be recruited. Sociodemographic and stroke-related variables (e.g., age, time since stroke) will be collected to confirm participant eligibility. Prior to training, participants will undergo a clinical evaluation of their affected UL as well as an evaluation of simulated pain at the affected UL. For the latter, the effect of CN-NINM on pain will be evaluated using a tonic thermal experimental pain paradigm. For this, a thermode (hot plate) will be applied to the forearm of the participants before and after a single 20-minute application of CN-NINM. On each occasion, thermal nociceptive stimuli will be induced for 2 minutes on the participants' forearm using the thermode. Although the temperature remains constant for the entire 2 minutes, the participant will be informed that the temperature may increase, decrease, or remain stable during the procedure. The participant will then, at all times, evaluate the intensity of the pain with a visual analogue scale connected to a computer (CoVAS: visual analogue scale from 0 to 100). Afterwards, the participants will take part in a 4-week training program of their affected UL (3X/week, 60-minute duration). During each training session, the CN-NINM will be applied for 20 minutes at an intensity tailored to each participant comfort.

ELIGIBILITY:
Inclusion Criteria:

1. Be ≥18 years old;
2. Have had a single supratentorial stroke;
3. Be in a chronic stroke phase (>6 months);
4. Present motor recovery in the upper limb (UL) (Fugl-Meyer Stroke Assessment [FMA] score ≥20/66);
5. Have completed any rehabilitation treatment.

Exclusion Criteria:

1. A significant spasticity at the affected upper limb (score > 3 on the modified Ashworth scale);
2. A major sensory deficit at the affected upper limb (a score ≤25/34 on the Nottingham Sensory Assessment and a score <6 on the evaluation of the vibration threshold);
3. A presence of hemineglect (score ≥±0. 083 on the Line Cancellation test);
4. An apraxia (score >2.5 on the Alexander Test);
5. The presence of a neurological disorder other than a stroke;
6. Concomitant orthopaedic problem at the affected UL;
7. Cognitive impairment (Mini-Cog score <2/5) and
8. Any contraindication to CN-NINM.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Actual)
Dates: Start 2022-06-27 (Actual); Primary Completion 2023-06-21 (Actual); Study Completion 2023-06-21 (Actual)

PRIMARY OUTCOMES:
Recruitment rate for the project | Information will be assessed at the end of the recruitment period, at week 28
  This outcome will be compiled by the total number of participants recruited, divided by the average number of months recruiting.
Refusal to participate and the reasons | Information will be assessed throughout the project recruitment period (average of 7 months)
  Participants refusal to participate will be assessed by number of participants who declined to participate in the project and the associate reasons
Dropped out rate of the project in percent and the reasons | Information will be assessed through project completion, an average of 9 months
  Dropped out rate will be collected by the number of participants who dropped out of the project divided by the total number of participants recruited X 100%. Reasons for each drop out will also be collected.
Adherence to the intervention (training program and CN-NINM) in percent | Information will be assessed through study completion, an average of 9 months
  Adherence to the intervention will be calculated by the number of training sessions completed out of the total number expected X 100%
Number of participants with CN-NINM-related adverse events as assessed by a questionnaire | Information will be be assessed through study completion, an average of 9 months
  Adverse events will be assessed with a questionnaire that will provide a number and percentage of participants who have experienced adverse events as well as allowing collecting information on symptoms that may be related to CN-NINM.

SECONDARY OUTCOMES:
Change in pain intensity on the CoVAS | The assessments will be done at the baseline and just after the 20 minutes of application of the CN-NINM.
  Change in pain intensity will be calculated by the difference between the pain felt and reported on the CoVAS (average of the 2 minutes) before and after the single application of CN-NINM. The score on the CoVAS ranges between 0 (no pain) to 100 (maximal pain).
Change in UL functional performance on the Wolf Motor Function Test | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in functional performance of the affected UL will be assessed with the timed score of the Wolf Motor Function Test; comprising 17 tasks. The maximal time allocated to each task is 120 seconds.
Change in UL motor function on the Fugl-Meyer Stroke Assessment Scale | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in motor function of the affected UL will be assessed using the Fugl-Meyer Stroke Assessment where a score of 66 is equivalent to full motor recovery.
Change in affected grip strength on the JAMAR dynamometer | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in affected grip strength will be assessed by computing the mean of 3 trials in kilograms on the JAMAR dynamometer.
Change in manual dexterity on the Box and Block test | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in manual dexterity will be assessed with the Box and Block Test, computing the number of blocks that can be transferred from one compartment to another in 60 seconds.
Change in participants' subjective real life functional UL performance on the Motor Activity Log | The assessments will be done at the baseline and in the week after completion of the training program and CN-NINM.
  Change in participants' self-reported affected UL performance in everyday activities will be assessed with the Motor Activity Log (MAL). The MAL comprises 14 task scored on a 0 to 5 Likert scale, where a score of 5 represents normal quantity and quality of use of affected UL.

CONTACTS AND LOCATIONS:
Overall Officials: Marie-Hélène Milot, Ph.D., Principal Investigator — Université de Sherbrooke; Guillaume Léonard, Ph.D., Principal Investigator — Université de Sherbrooke
Locations (1):
- Centre de recherche sur le vieillissement, Sherbrooke, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No
The investigators are not planning on sharing individual data to the participants.

REFERENCES:
- [Derived] Ahiatsi M, Milot MH, Flaive A, Leonard G. Tasting pain-relief through tongue stimulation: results from a feasibility study looking into the use of cranial nerve non-invasive neuromodulation in healthy individuals and chronic poststroke patients. BMC Neurol. 2026 Jan 2. doi: 10.1186/s12883-025-04498-6. Online ahead of print. PMID 41484860
- [Derived] Ahiatsi M, Leonard G, Riesco E, Girard MC, Milot MH. A feasibility study on the use of cranial nerve non-invasive neuromodulation to improve affected arm function in people in the chronic stage of a stroke. BMC Neurol. 2025 May 16;25(1):208. doi: 10.1186/s12883-025-04213-5. PMID 40380081